CLINICAL TRIAL: NCT01879241
Title: Efficacy, Safety and Tolerability Study of 1 mg Rasagiline in Patients With Amyotrophic Lateral Sclerosis (ALS) Receiving Standard Therapy (Riluzole) - An AMG Trial With a Market Authorized Substance
Brief Title: Study of Rasagiline in Patients With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Albert Christian Ludolph, Prof., MD, Prof., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAS-ALS; 2011-004482-32 (EudraCT Number)
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; survival time; ALS functioning Rating Scale; quality of life; survival
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rasagiline (Experimental): Rasagiline
  1 mg/day; 18 months
  Interventions: Drug: Rasagiline
- Placebo (Placebo Comparator): once daily, 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasagiline
  Arms: Rasagiline
Drug: Placebo — a sugar pill manufactured to mimic Rasagiline 1 mg tablet
  Arms: Placebo

SUMMARY:
The primary objective of the trial is to investigate the survival time (the time from randomization until death or end of the trial) compared between control group and experimental group.

This is a prospective, multicenter, randomized, stratified, parallel-group, double-blind trial comparing placebo with 1 mg/d rasagiline as add-on therapy to 100 mg riluzole in amyotrophic lateral sclerosis (ALS) in 250 enrolled patients. For entry, the El Escorial Criteria for the diagnosis of ALS will be used. The patients have to be stable on riluzole at least 4 weeks prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Possible, probable (clinically or laboratory) or definite ALS according to the revised version of the El Escorial World Federation of Neurology criteria
* Disease duration more than 6 months and less than 3 years (inclusive). Disease onset defined as date of first muscle weakness, excluding fasciculations and cramps
* Vital capacity more than 50% of normal (slow vital capacity; best of three measurements)
* Age: ≥ 18 years
* Continuously treated with 100 mg riluzole for at least four weeks
* Capable of thoroughly understanding all information given and giving full informed consent according to GCP
* Women of childbearing age must be non-lactating and surgically sterile or using a highly effective method of birth control and have a negative pregnancy test. Acceptable methods of birth control with a low failure rate i.e. less than 1% per year) when used consistently and correct are such as implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), or double-barrier methods (condom or diaphragm with spermicidal agent or IUD), sexual abstinence or vasectomized partner

Exclusion Criteria:

* Previous participation in another clinical study within the preceding 12 weeks
* Tracheostomy or assisted ventilation of any type during the preceding three months
* Gastrostomy
* Any medical condition known to have an association with motor neuron dysfunction which might confound or obscure the diagnosis of ALS
* Presence of any concomitant life-threatening disease or impairment likely to interfere with functional assessment
* Patients on sympathomimetic agents. This includes pseudoephedrine, phenylephrine, phenylpropanolamine, and ephedrine.
* Patients on analgesics with serotoninergic properties such as meperidine, tramadol, methadone and propoxyphene.
* Patients on serotonin reuptake inhibitors (SSRIs). This includes fluoxetine or fluvoxamine.
* Patients on dextromethorphan, St. John's wort, cyclobenzaprine or other MAO inhibitors (selective or non-selective)
* Patients taking Antidepressants
* Confirmed hepatic insufficiency or abnormal liver function (ASAT and/or ALAT greater than 3 times the upper limit of the normal range)
* Renal insufficiency (serum creatinine more than 2.26 mg/dL)
* Evidence of major psychiatric disorder or clinically evident dementia precluding evaluation of symptoms
* Known hypersensitivity to any component of the study drug
* Liable to be not cooperative or comply with the trial requirements (as assessed by the investigator), or unable to be reached in the case of emergency
* Female with childbearing potential, if no adequate contraceptive measures are used
* Pregnancy or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Survival in ALS-Patients with Rasagiline compared to placebo | 18 Months

SECONDARY OUTCOMES:
Change of total score of ALS Functional Rating Scale - Revised (ALSFRS-R) | 18 Months
Change of individual Quality of Life (SEIQoL, Schedule for the Evaluation of Individual Quality of Life | 18 Months
Change of slow vital capacity | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Albert C. Ludolph, MD, Prof., Principal Investigator — Department of Neurology, University of Ulm
Locations (15):
- Germany (15):
  - Department of Neurology, University of Ulm, Ulm, Baden-Wurttemberg
  - Department of Neurology, Technische Universität München, Munich, Bavaria
  - Department of Neurology, Universty of Regensburg, Regensburg, Bavaria
  - Department of Neurology, University of Wuerzburg, Würzburg, Bavaria
  - Department of Neurology, Deutsche Klinik für Diagnostik, Wiesbaden, Hesse
  - Department of Neurology, University of Goettingen, Göttingen, Lower Saxony
  - Department of Neurology, Medical School Hannover, Hanover, Lower Saxony
  - Department of Neurology, University of Rostock, Rostock, Mecklenburg-Vorpommern
  - Department of Neurology, Universty of Bonn, Bonn, Nordrhrein-Westfalen
  - Neurologische Universitätsklinik Bergmannsheil, Bochum, North Rhine-Westphalia
  - Department of Neurology, Universty of Muenster, Münster, North Rhine-Westphalia
  - Department of Neurology, TU Dresden, Dresden, Saxony
  - Department of Neurology, University of Halle-Wittenberg, Halle, Saxony-Anhalt
  - Department of Neurology, University of Jena, Jena, Thuringia
  - Department of Neurology, Humboldt University, Berlin

REFERENCES:
- [Background] Waibel S, Reuter A, Malessa S, Blaugrund E, Ludolph AC. Rasagiline alone and in combination with riluzole prolongs survival in an ALS mouse model. J Neurol. 2004 Sep;251(9):1080-4. doi: 10.1007/s00415-004-0481-5. PMID 15372249
- [Derived] Ludolph AC, Schuster J, Dorst J, Dupuis L, Dreyhaupt J, Weishaupt JH, Kassubek J, Weiland U, Petri S, Meyer T, Grosskreutz J, Schrank B, Boentert M, Emmer A, Hermann A, Zeller D, Prudlo J, Winkler AS, Grehl T, Heneka MT, Wollebaek Johannesen S, Goricke B; RAS-ALS Study Group. Safety and efficacy of rasagiline as an add-on therapy to riluzole in patients with amyotrophic lateral sclerosis: a randomised, double-blind, parallel-group, placebo-controlled, phase 2 trial. Lancet Neurol. 2018 Aug;17(8):681-688. doi: 10.1016/S1474-4422(18)30176-5. Epub 2018 Jun 19. PMID 29934198